CLINICAL TRIAL: NCT03484442
Title: Role of Multislice Computed Tomography Angiography In Diagnosis oF Clinically Suspected Acute Mesenteric Ischemia
Brief Title: Multislice Computed Tomography Angiography in Acute Mesenteric Ischemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Basma Fawzy Mohammed, principle investigator, Assiut University
Other Study IDs: CTA
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Mesenteric Ischemia
MeSH Terms: conditions — Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute mesenteric ischemia is a life-threatening condition with high mortality. Acute mesenteric ischemia is responsible for fewer than one in 1000 hospital admissions, but its mortality rate ranges between 30% and 90% . Acute mesenteric ischemia is most commonly secondary to embolism followed by arterial thrombosis, non-occlusive ischemia, and less commonly venous thrombosis . Delay in diagnosis contributes to the continued high mortality rate. Early diagnosis and prompt effective treatment are essential to Correspondence to improve clinical outcomes

DETAILED DESCRIPTION:
However, Acute mesenteric ischemia represents a major diagnostic challenge because of its varied presentations and multiple causes . Patients usually present with non-specific abdominal symptoms and laboratory findings, which leads to delayed diagnoses . Therefore, diagnostic imaging has emerged as one of the most crucial components in the diagnostic work-up of suspected

Recent technical advances have made computed tomography angiography the modality of choice in the setting of suspected Acute mesenteric ischemia.computed tomography angiography is a rapid and non-invasive diagnostic tool for assessing intestinal vasculature and bowel . computed tomography angiography allows early diagnosis and differentiation between occlusive and non-occlusive causes, which is important to direct therapeutic approach . Overall, combining vascular and bowel assessment results in a high diagnostic accuracy . A recent meta-analysis showed a sensitivity of 93% and a specificity of 96% . However, this meta analysis also showed that the prevalence of confirmed .Acute mesenteric ischemia is less than 25% among the patients referred to computed tomography angiograph in the setting of suspected Acute mesenteric ischemia .Knowledge of the prevalence and the demographic distribution of alternative diagnoses in the remaining three-fourths of patients without Acute mesenteric ischemia is important for appropriate patient care. computed tomography angiograph is considered to allow for a variety of acute alternative diagnoses, ensuring timely triage of these patients.

ELIGIBILITY:
Inclusion Criteria:

Clinically suspected acute mesenteric ischemia based on physician evaluation Patients should be evaluated during 48 h of acute presentation

Exclusion Criteria:

* Renal Impairment
* Known allergy to iodine contrast media.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinically suspected acute mesentric ischemia based on physician evaluation Patients should be evaluated during 48 h of acute presentation
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
rate of diagnosis of Acute mesenteric ischemia | 48 hours of presentation
  number of patients accurately diagnosed acute mesenteric ischemia by multislice computed tomography angiography

REFERENCES:
- [Background] Ottinger LW. Mesenteric ischemia. N Engl J Med. 1982 Aug 26;307(9):535-7. doi: 10.1056/NEJM198208263070905. No abstract available. PMID 7048095
- [Background] Ozden N, Gurses B. Mesenteric ischemia in the elderly. Clin Geriatr Med. 2007 Nov;23(4):871-87, vii-viii. doi: 10.1016/j.cger.2007.07.001. PMID 17923343
- [Background] Herbert GS, Steele SR. Acute and chronic mesenteric ischemia. Surg Clin North Am. 2007 Oct;87(5):1115-34, ix. doi: 10.1016/j.suc.2007.07.016. PMID 17936478
- [Background] Paterno F, Longo WE. The etiology and pathogenesis of vascular disorders of the intestine. Radiol Clin North Am. 2008 Sep;46(5):877-85, v. doi: 10.1016/j.rcl.2008.06.005. PMID 19103137
- [Background] Reginelli A, Iacobellis F, Berritto D, Gagliardi G, Di Grezia G, Rossi M, Fonio P, Grassi R. Mesenteric ischemia: the importance of differential diagnosis for the surgeon. BMC Surg. 2013;13 Suppl 2(Suppl 2):S51. doi: 10.1186/1471-2482-13-S2-S51. Epub 2013 Oct 8. PMID 24267670
- [Background] Cudnik MT, Darbha S, Jones J, Macedo J, Stockton SW, Hiestand BC. The diagnosis of acute mesenteric ischemia: A systematic review and meta-analysis. Acad Emerg Med. 2013 Nov;20(11):1087-100. doi: 10.1111/acem.12254. PMID 24238311
- [Background] Martinez JP, Hogan GJ. Mesenteric ischemia. Emerg Med Clin North Am. 2004 Nov;22(4):909-28. doi: 10.1016/j.emc.2004.05.002. PMID 15474776
- [Background] Sise MJ. Acute mesenteric ischemia. Surg Clin North Am. 2014 Feb;94(1):165-81. doi: 10.1016/j.suc.2013.10.012. PMID 24267504
- [Background] Ofer A, Abadi S, Nitecki S, Karram T, Kogan I, Leiderman M, Shmulevsky P, Israelit S, Engel A. Multidetector CT angiography in the evaluation of acute mesenteric ischemia. Eur Radiol. 2009 Jan;19(1):24-30. doi: 10.1007/s00330-008-1124-5. Epub 2008 Aug 9. PMID 18690454
- [Background] Menke J. Diagnostic accuracy of multidetector CT in acute mesenteric ischemia: systematic review and meta-analysis. Radiology. 2010 Jul;256(1):93-101. doi: 10.1148/radiol.10091938. PMID 20574087